CLINICAL TRIAL: NCT03244007
Title: Evaluation of Retinal Microstructure Detected With Intraoperative Optical Coherence Tomography During Vitrectomy
Status: Completed | Type: Observational
Sponsor: Kyorin University (Other)
Responsible Party: Principal Investigator, Makoto Inoue, Professor of Ophthalmology, Kyorin University
Other Study IDs: Kyorineye023
Record Dates: First submitted 2017-08-05; First posted 2017-08-09 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Macular Disease
Keywords: macular hole; lamellar macular hole
MeSH Terms: conditions — Macular Degeneration; Retinal Perforations | interventions — Vitrectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Eyes with residual fragment: The eyes with residual fragments detected with intraoperative optical coherence tomography
  Interventions: Procedure: Vitrectomy
- Eyes without residual fragment: The eyes without residual fragments detected with intraoperative optical coherence tomography
  Interventions: Procedure: Vitrectomy

INTERVENTIONS:
Procedure: Vitrectomy

SUMMARY:
We evaluate the intraoperative optical coherence tomographic (OCT) images of eyes with idiopathic macular hole (MH) or lamellar macular hole whether the intraoperative OCT findings will affect postoperative visual outcome.

DETAILED DESCRIPTION:
We evaluate the intraoperative optical coherence tomographic (OCT) images of eyes with idiopathic macular hole (MH) or lamellar macular hole whether the intraoperative OCT findings will affect postoperative visual outcome.

ELIGIBILITY:
Inclusion Criteria: Eyes with macular hole or lamellar macular hole -

Exclusion Criteria: Eyes with retinal detachment, retinal vascular disease, glaucoma

-

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The eyes with macular hole or lamellar macular hole
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-12-12 (Actual); Primary Completion 2016-12-11 (Actual); Study Completion 2017-06-11 (Actual)

PRIMARY OUTCOMES:
Recovery of microstructure | 6 months

SECONDARY OUTCOMES:
Visual improvement | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Inoue, MD, Principal Investigator — Korin Eye Center
Locations (1):
- Makoto Inoue, Mitaka-shi, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No